CLINICAL TRIAL: NCT06504238
Title: Non-Invasive Monitoring Methods in Patients With Acute Brain Injury
Acronym: NIMABI
Status: Recruiting | Type: Observational
Sponsor: Boston Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: H-44955
Record Dates: First submitted 2024-07-09; First posted 2024-07-16 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: Brain Injury, Acute
Keywords: Life-threatening mass effect (LIME); Traumatic brain injury (TBI); Ischemic stroke (IS); Intraparenchymal hemorrhage (IPH); Neurologic deterioration; Intracranial Pressure (ICP); Glasgow Coma Scores
MeSH Terms: conditions — Brain Injuries; Brain Injuries, Traumatic; Ischemic Stroke

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — The investigators are building a repository of demographic, invasive ICP monitoring data, clinical, laboratory, diagnostic, treatment (medical and surgical) and outcome data will be collected (variables below). Data will be collected from non-invasive devices using either clinical review from the chart, or if not available and/or used for additional measurements, from the device (smartguard for pupillometry, imaging, EEG data, Brain4care data). The limited dataset (the only identifiers being dates of pupil measurements/medical services) will be maintained in a password secured and HIPAA protected REDCap database.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- NIMABI Group: Eligible patients will be recruited on admission to the ICU followed by the Neurointensive care team.
  Demographic, invasive ICP monitoring data, clinical, laboratory, diagnostic, treatment (medical and surgical) and outcome data will be collected. Data will be collected from non-invasive devices using either clinical review from the chart, or if not available and/or used for additional measurements, from the device (smartguard for pupillometry, imaging, EEG data, Brain4care data).

SUMMARY:
Life-threatening mass effect (LTME) arises when brain swelling displaces or compresses crucial midline structures subsequent to acute brain injuries (ABIs) like traumatic brain injury (TBI), ischemic stroke (IS), and intraparenchymal hemorrhage (IPH), which can manifest rapidly within hours or more gradually over days. Despite advancements in surgical management, significant gaps in understanding persist regarding optimal monitoring and therapeutic approaches. The current standard for identifying LTME involves neurologic decline in conjunction with radiographic evidence or increased intracranial pressure (ICP) indicating space-occupying mass effect. However, in critically ill patients, reliance on subjective physical exam findings, such as decreased arousal, often leads to delayed recognition, occurring only after catastrophic shifts have already occurred.

The goal of this study is to determine the association of non-invasive biomarkers with neurologic deterioration, and to determine whether non-invasive biomarker inclusion improves detection of outcome and decline.

The investigators propose to use various non-invasive methods to monitor ICP as adjuncts in detecting deteriorating mass effect. These methods include quantitative pupillometry, radiographic data, laboratory data, and other bedside diagnostic tests available including electroencephalography (EEG), skull vibrations detected via brain4care device, optic nerve sheath diameter assessment (ONSD), and ultrasound-guided eyeball compression. Some of these methods will be measured *only* for the purposes of the research study (such as skull vibrations via brain4care). Other measurements, such as quantitative pupillometry, will represent additional measurements beyond those already being collected for clinical care. This research study is necessary to understand the association of these non-invasive biomarkers with neurological decline and outcomes while considering potential confounding factors.

ELIGIBILITY:
Inclusion Criteria:

* Admitted under Neuro intensivist primary or consultative care.
* At least one head computed tomography (CT) scan demonstrating intracranial pathology that may lead to life-threatening mass effect (i.e. traumatic brain injury, ischemic or hemorrhagic stroke, epidural or subdural hematoma, subarachnoid hemorrhage, diffuse hypoxic injury, metabolic cerebral edema, tumor)
* Concern for Life Threatening Mass Effect
* Glasgow Coma Score (GCS) <9
* Anticipated stay >24 hours

Exclusion Criteria:

* Comfort measure only
* Any other criteria that the PI deems that makes the patient inadequate for the study
* Sub-exclusion criteria for specific non-invasive measurements include:

  * Orbital injury (pupillometry, ONSD)
  * Traumatic injury or surgery that precludes use of B4C device
* Presence of supratentorial craniectomy or craniotomy that has not healed and is mobile/bone defects/scalp injury [EEGelectroencephalogram (EEG), Brain4Care]
* Presence of extensive scalp injury

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible patients will be recruited on admission to the intensive care unit (ICU) at Boston Medica Center followed by the Neurointensive care team.
Sampling Method: Non-Probability Sample
Enrollment: 720 (Estimated)
Dates: Start 2024-09-26 (Actual); Primary Completion 2030-09 (Estimated); Study Completion 2030-09 (Estimated)

PRIMARY OUTCOMES:
Neurologic Deterioration | 5 years
  Neurologic deterioration will be assessed as a dichotomous variable (yes/no) defined as a negative change in any of the following: level of consciousness, agaze, arm motor function, leg motor function, or language. The participants' medical chart will be reviewed for documentation of persistent change.
Glasgow Coma Scores | 5 years
  The Glasgow Coma Scale (GCS) is a 15-point scale used to evaluate a person's state of consciousness. A score of 3 is the lowest possible and indicates a deep coma or death, while a score of 15 is the highest and indicates a fully awake person. A lower score generally means a deeper coma.

SECONDARY OUTCOMES:
Number of participant deaths during hospitalization | 5 years
  This data will be abstracted from medical records..
Functional outcome at hospital discharge | 5 years
  This will be assessed by Modified Rankin Scale (mRS), a 6 point disability scale with possible scores ranging from 0 to 5, higher scores indicating greater disability and where 0-2 is generally considered a good outcome with individuals assuming complete functional independence. A separate category of 6 is usually added for patients who expire. Data will be abstracted from medical records on review of patient notes and discharge summaries to obtain amRS for each participant.

CONTACTS AND LOCATIONS:
Overall Officials: Charlene Ong, MD MPHS, Principal Investigator — Boston Medical Center, Neurology
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No